CLINICAL TRIAL: NCT05477212
Title: Evaluation of Gut Permeability in Patients Affected by Obesity and NAFLD: Influence of Ketogenic Diet on Diagnostic and Prognostic Markers in Liver Disease
Brief Title: Evaluation of Gut Permeability in Patients Affected by Obesity and NAFLD: Influence of Ketogenic Diet.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Collaborators: Francesco Russo (Unknown); Giuseppe, Riezzo (Unknown); Michele, Linsalata (Unknown); Antonella, Orlando (Unknown); Benedetta, D Attoma (Unknown); Laura, Prospero (Unknown); Antonia, Ignazzi (Unknown); Sara, De Nucci (Unknown); Raffaele, Cozzolongo (Unknown); Vito, Giannuzzi (Unknown); Maria, De Angelis (Unknown); Giusy Rita, Caponio (Unknown); Oronzo, Milella (Unknown); Gianluigi, Giannelli (Unknown)
Responsible Party: Principal Investigator, Prof. Giovanni De Pergola, MD, Professor, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NAFLDdietachetogenica
Record Dates: First submitted 2022-07-18; First posted 2022-07-28 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Permeability; Increased; NAFLD; Obesity
Keywords: obesity; Gut permeability; NAFLD; Ketogenic diet
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention arm with VLCKD (Experimental): all patients will receive a very low calorie Ketogenic diet (VLCKD) and will be followed for all the time of the study, monitoring gut permeability, liver steatosis and microbiome composition
  Interventions: Dietary Supplement: Ketogenic Diet

INTERVENTIONS:
Dietary Supplement: Ketogenic Diet — all patients will receive a very low calorie ketogenic diet

SUMMARY:
This study is open label, with one arm only. In this study will be enrolled patients with obesity (BMI more than 30). Aim of the study is to determine the influence (if any) of a very low calorie ketogenic diet (VLCKD) on gut permeability and liver steatosis.

The first objective is to examine the influence of obesity on the prevalence and severity of impaired intestinal permeability and hepatic steatosis.

Intestinal permeability means the ability of the intestinal barrier to block the passage of substances potentially harmful to our body.

The second objective is to evaluate whether a low-calorie and ketogenic dietary intervention, lasting 6 weeks, can change intestinal permeability and hepatic steatosis

ELIGIBILITY:
Inclusion Criteria:

1. BMI ≥ 30 Kg/m2 or abdominal circumference (waist) >94 cm in men and >80 cm in women (IDF criteria for the definition of abdominal obesity) with or without the features that characterize the metabolic syndrome
2. Age range between 18 and 70 years, both sexes
3. Diagnosis of hepatic steatosis, formulated on the basis of fibroscan [CAP (controlled attenuation parameter) > 238 dB/m(decibel/meter)], and other recognized criteria (FLI - Fatty Liver Index , FIB-4 - Fibrosis-4 index, NFS - NAFLD fibrosis score).

Exclusion Criteria:

1. Normal and underweight subjects
2. Presence of any pathology that may affect the presence of altered intestinal permeability or steatosis, apart from pathologies that represent inclusion criteria
3. Treatment with any device, pharmacological or not, that can affect intestinal permeability and liver metabolism and, therefore, the presence of steatosis
4. Pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2025-05-28 (Estimated)

PRIMARY OUTCOMES:
Gut permeability | 6 weeks
  examine the influence of obesity on possible alterations (if any) in intestinal permeability. subjects drank a sugar test solution containing 10 g of lactulose, 5 g of mannitol, and 40 g of sucrose in a volume of 100 ml. Urine samples were collected up to 5 h after administration. . Te percentage of ingested La (%La), Ma (%Ma), and Su (%Su) were evaluated in urine, and the La/Ma ratio was calculated for each sample. Patients with a La/Ma ratio higher than 0.030 were considered as having an altered gut permeability
Gut Dysbiosis | 6 weeks
  evaluate the impact of the low-calorie and ketogenic diet on possible alterations of the intestinal microbiome.
  The dysbiosis test is based on urinary quantification of two metabolites deriving from the decomposition of tryptophan, skatole (3-methyl-indole), and indican.
  Urinary indican and skatole were considered normal at values lower than 10 mg/L and 10 µg/L, respectively. Urinary concentrations of indican and skatole higher than 20 mg/L and 20 µg/L indicate the presence of fermentative and putrefactive grade I dysbiosis, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni De Pergola, Prof, Principal Investigator — IRCCS "Saverio de Bellis"
Locations (1):
- Irccs Saverio de Bellis, Castellana Grotte, BARI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Genser L, Aguanno D, Soula HA, Dong L, Trystram L, Assmann K, Salem JE, Vaillant JC, Oppert JM, Laugerette F, Michalski MC, Wind P, Rousset M, Brot-Laroche E, Leturque A, Clement K, Thenet S, Poitou C. Increased jejunal permeability in human obesity is revealed by a lipid challenge and is linked to inflammation and type 2 diabetes. J Pathol. 2018 Oct;246(2):217-230. doi: 10.1002/path.5134. Epub 2018 Aug 28. PMID 29984492
- [Result] Damms-Machado A, Louis S, Schnitzer A, Volynets V, Rings A, Basrai M, Bischoff SC. Gut permeability is related to body weight, fatty liver disease, and insulin resistance in obese individuals undergoing weight reduction. Am J Clin Nutr. 2017 Jan;105(1):127-135. doi: 10.3945/ajcn.116.131110. Epub 2016 Nov 9. PMID 28049662
- [Result] Mkumbuzi L, Mfengu MMO, Engwa GA, Sewani-Rusike CR. Insulin Resistance is Associated with Gut Permeability Without the Direct Influence of Obesity in Young Adults. Diabetes Metab Syndr Obes. 2020 Aug 24;13:2997-3008. doi: 10.2147/DMSO.S256864. eCollection 2020. PMID 32922055
- [Result] Ott B, Skurk T, Hastreiter L, Lagkouvardos I, Fischer S, Buttner J, Kellerer T, Clavel T, Rychlik M, Haller D, Hauner H. Effect of caloric restriction on gut permeability, inflammation markers, and fecal microbiota in obese women. Sci Rep. 2017 Sep 20;7(1):11955. doi: 10.1038/s41598-017-12109-9. PMID 28931850
- [Result] Muscogiuri G, El Ghoch M, Colao A, Hassapidou M, Yumuk V, Busetto L; Obesity Management Task Force (OMTF) of the European Association for the Study of Obesity (EASO). European Guidelines for Obesity Management in Adults with a Very Low-Calorie Ketogenic Diet: A Systematic Review and Meta-Analysis. Obes Facts. 2021;14(2):222-245. doi: 10.1159/000515381. Epub 2021 Apr 21. PMID 33882506